CLINICAL TRIAL: NCT05482607
Title: Unsupervised Clustering Evaluation of HRCT Patterns in Systemic Sclerosis-associated Interstitial Lung Disease
Brief Title: Evaluation of HRCT Patterns in Systemic Sclerosis-associated Interstitial Lung Disease
Acronym: LUNGSCLEROCT
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI105
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SSc-ILD patients

SUMMARY:
Systemic sclerosis (SSc) is a heterogeneous systemic autoimmune disease with distinct prognosis according to patients. Interstitial lung disease (ILD) concerns almost 50 % of SSc patients and represents the main cause of mortality. SSc-ILD is variable: from limited forms (with asymptomatic patients) to extensive lesions. Disease course in SSc-ILD is also highly variable: patients can experience stable disease, slow or fast progression. Investigators performed unsupervised clustering analysis to classify SSc-ILD according to elementary radiological lesions on HRCT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis according to 2013 ACR/EULAR criteria
* Patients with interstitial lung disease on HRCT chest

Exclusion Criteria:

* Patients with an alternative diagnosis of SSc-associated ILD (silicosis, sarcoidosis, lung cancer or other significant lung abnormalities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis-interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
HRCT scan variables | baseline (J0)
  HRCT scan variables included in hierarchical agglomerative clustering (HAC) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Decker, MD, Principal Investigator — CHU NANCY
Locations (1):
- Central Hospital, Nancy, France